CLINICAL TRIAL: NCT01181687
Title: Psychometric Testing of the Norwegian Version of the Comfort Behavioral Scale
Status: Completed | Type: Observational
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Geir Hoff, Professor, Sykehuset Telemark
Other Study IDs: 2010/1268 (REK)
Record Dates: First submitted 2010-08-03; First posted 2010-08-13 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Postoperative Pain
Keywords: COMFORT behavioral scale; pain assessment scale; child; validity; reliability
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to establish reliability and validity of the Norwegian version of the Comfort behavioral scale.

DETAILED DESCRIPTION:
Structured pain assessment is the foundation for the management of pain. Several different pain measurement tools exists, among them the Comfort behavioral scale (van Dijk, 2005), developed from the original Comfort scale (Ambuel, 1992). The psychometric properties of the Comfort scale have been tested in several studies, but so far no Norwegian version of the scale has been developed and tested. Neither has the scale been tested in spontaneously breathing children undergoing minor surgery. The aim of this study is to establish incipient psychometric properties of the Norwegian version of the scale among children aged 0-3 years admitted for elective minor surgery.

ELIGIBILITY:
Inclusion Criteria:

* Younger than 3 years old at the time of surgery
* Day care patients admitted for minor elective surgery

Exclusion Criteria:

* Pre-entry use of sedation and/or analgesics
* Neurological or other diseases or drugs (neuromuscular blockers) thet significantly influence motor activity, facial expression, cognition, or emotional state, ex. cerebral palsy, myopathy, severe mental retardation, severe hypotonia, neuromuscular disease

Ages: 40 Weeks to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children admitted to Telemark Hospital (level II hospital) and meeting the inclusion and exclusion criteria specified
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Increase in Comfort behavioral scale score | Within 24 hours after admission to the hospital for surgery
  Testing the hypothesis that there will be a clincal significant increase in Comfort-score when the scores from admission and after surgery are compared. The highest registered score obtained during the first 24 hours after surgery will be used for this analysis. We assume that the score at admission reflects no pain/sedation, while the scores after surgery reflect varying degree of pain

SECONDARY OUTCOMES:
Convergent validity of the Comfort behavioral scale | Within 24 hours after admission to the hospital for surgery
  The correlations between each of the items of the scale and between each item and the overall Comfort behavioral scale-score will be calculated
Inter-rater reliability of the Comfort behavioral scale | Within 24 hours after admission to the hospital for surgery
  Calculate the inter-rater reliability among nurses for the Norwegian version of the Comfort behavioral scale
Reduction in Comfort behavioral scale score (2) | Within 24 hours after admission to the hospital for surgery
  Testing the hypothesis that there will be a clinically significant reduction in Comfort-score when the scores from after the administration of pre-medication and after surgery when the child still has a laryngeal mask in place is compared. We assume that the score after premedication is given reflects a light sedation while the scores after surgery when the child still has a laryngela mask in place reflects deep sedation.
Reduction in Comfort behavioral scale score (1) | Within 24 hours after admission to the hospital for surgery
  Testing the hypothesis that there will be a clincal significant reduction in Comfort-score when the scores from admission and after the administration of pre-medication are compared. We assume that the score at admission reflect no pain/sedation, while the scores after pre-medication is given reflect sedation

CONTACTS AND LOCATIONS:
Overall Officials: Leena Jylli, PhD, Study Chair — Karolinska Institutet
Locations (1):
- Telemark Hospital, Skien, Telemark, Norway